CLINICAL TRIAL: NCT06277921
Title: 90-day Postoperative Morbidity and Mortality After Elective Surgery for Esophageal and Esophagogastric Junction Cancer
Brief Title: Morbidity and Mortality After Esophageal and Esophagogastric Junction Cancer Surgery
Acronym: ESOSTAT
Status: Completed | Type: Observational
Sponsor: P. Herzen Moscow Oncology Research Institute (Other Government)
Collaborators: National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Principal Investigator, Andrey Ryabov, Head of Department of Thoracoabdominal Oncology, P. Herzen Moscow Oncology Research Institute
Other Study IDs: 110-2
Record Dates: First submitted 2024-02-08; First posted 2024-02-26 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer; Oesophageal Cancer; Siewert Type I Adenocarcinoma of Esophagogastric Junction; Siewert Type III Adenocarcinoma of Esophagogastric Junction
Keywords: Esophageal Cancer; Esophagogastric Junction Cancer; Morbidity; Mortality; Surgery
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with morbidity and mortality: Patients who suffered from any type of morbidity after surgery
  Interventions: Procedure: Elective Surgery for gastric cancer
- Patients without morbidity and mortality: Patients who did not suffer from any type of morbidity after surgery
  Interventions: Procedure: Elective Surgery for gastric cancer

INTERVENTIONS:
Procedure: Elective Surgery for gastric cancer — Resection of the esophagus and the gastroesophageal junction via open, laparoscopic or robotic approach
  Other Names: Esophageal or Esophagogastric Junction Cancer

SUMMARY:
Esophageal and esophagogastric junction cancer is still one of the main health care issue and esophagectomy with lymph node dissection is the only chance to be cure.

However, esophagectomy for esophageal cancer is a complex procedure which carries high risk of morbidity rate of 24% and a mortality rate of 2% to 5.6%, respectively There is a need to study the differences of 90-day postoperative morbidity and mortality in different clinics and centers of the Russian Federation.

DETAILED DESCRIPTION:
Esophageal and esophago-gastric junction cancer is the seventh most common malignancy and the sixth leading cause of cancer-related mortality worldwide.

Surgery remains the primary treatment for esophageal cancer and is one of the most technically challenging interventions in oncological surgery. In addition, esophagectomy is associated with high risks of postoperative complications, with rates varying from clinic to clinic. Esophagectomy for esophageal cancer is a complex procedure which carries high risk of morbidity rate of 24% and a mortality rate of 2% to 5.6%, respectively.

The problem with the available studies of the course of the postoperative period is the significant heterogeneity of research methods, which does not allow us to obtain a true picture of the results of surgical treatment of the esophagus and esophagogastric junction cancer in the Russian Federation.

To improve the quality of further studies and recommendations on standardization of surgical treatment of esophageal and esophagogastric junction cancer and its morbidity, there is a need to study the differences of 90-day postoperative morbidity and mortality in different clinics and centers of the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with clinically documented primary Esophageal or Esophagogastric Junction malignancy (including Siewert I and II) undergoing elective surgery with curative intent - via open, laparoscopic or robotic approach between 18th March 2024 and 18th September 2024

Exclusion Criteria:

* Patients with clinical evidence of metastatic disease, including positive peritoneal cytology on a previous staging laparoscopy, or those with known synchronous other cancers.
* Esophagogastric Junction Siewert III malignancy
* Patients submitted to Emergency surgery or surgery without curative intent
* Patients undergoing any other surgery in addition to the curative surgery for primary Esophageal or Esophagogastric Junction malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with clinically documented primary Esophageal or Esophagogastric Junction malignancy (including Siewert I and II) undergoing elective surgery with curative intent - via open, laparoscopic or robotic approach
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
the type of complications and the incidence of it | within 90 days after operation
  the types of complication is classified into as follows: gastrointestinal (anastomotic leak, conduit necrosis/failure, pancreatitis, GI Bleeding, delayed conduit emptying); pulmonary (pneumonia, pleural effusion, pneumothorax, respiratory failure, ARDS, acute aspiration, tracheobronchial Injury); cardiac; thromboembolic; urologic; infection (wound infection; intrathoracic/intra-abdominal abscess; generalized sepsis; other infections); neurologic (recurrent nerve injury, acute delirium) and other (thoracic wound dehiscence, diaphragmatic hernia, chyle leak, reoperation other than for anastomotic leak or conduit necrosis, multiple organ dysfunction syndrome) complications Each complication will be graded according to Clavien-Dindo classification. Re-admission or visiting emergency room will be checked and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Ryabov, MD, PhD, Study Director — P.Herzen Moscow Oncological Research Institute; Vladimir Khomyakov, MD, PhD, Principal Investigator — P.Herzen Moscow Oncological Research Institute; Nuriddin Abdulkhakimov, MD, PhD, Principal Investigator — P.Herzen Moscow Oncological Research Institute; Pavel Smirnov, Principal Investigator — P.Herzen Moscow Oncological Research Institute
Locations (18):
- N.Alexandrov National Cancer Centre of Belarus, Minsk, Belarus
- Russia (17):
  - Bryansk Regional Oncological Hospital, Bryansk
  - Cheboksary Republican Clinical Oncology Dispensary, Cheboksary
  - M.Sigal Republican Medical Oncology Dispensary, Kazan'
  - A.Loginov Moscow Clinical Scientific Center, Moscow
  - Moscow City Oncology Hospital № 62, Moscow
  - P.Herzen Moscow Oncological Research Institute, Moscow
  - S.Yudin Moscow Oncological Center No.1, Moscow
  - University Clinical Hospital №1 of Sechenov University, Moscow
  - University Clinical Hospital №4 of Sechenov University, Moscow
  - Vishnevsky National Medical Research Center of Surgery, Moscow
  - Nizhny Novgorod Regional Clinical Oncological Dispensary, Nizhny Novgorod
  - Novosibirsk Regional Clinical Oncology Dispensary, Novosibirsk
  - A.Tsyb Medical Radiological Research Centre, Obninsk
  - Rostov-on-Don National Medical Research Centre for Oncology, Rostov-on-Don
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Saratov Regional Clinical Oncological Dispensary, Saratov
  - Ufa Republican Clinical Oncology Dispensary, Ufa